CLINICAL TRIAL: NCT04374591
Title: The Role of Sodium Bicarbonate as Adjuvant Treatment of Computed Tomography Identified COVID-19 Pneumonia: A Preliminary Report of Short Term Follow up
Brief Title: The Role of Sodium Bicarbonate as Adjuvant Treatment of Computed Tomography Identified COVID-19 Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sodium Bicarbonate COVID-19
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-07

CONDITIONS: Pneumonia; Covid19
Keywords: COVID-19
MeSH Terms: conditions — Pneumonia; COVID-19 | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate (Other): Inhalation of Sodium Bicarbonate 8.4% via nebulizer
  Interventions: Drug: Sodium Bicarbonate
- Control (Placebo Comparator): placebo
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium Bicarbonate — Inhalation of Sodium Bicarbonate 8.4% via nebulizer

SUMMARY:
To report the possible role of S.B 8.4% in the treatment of COVID-19pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Fever ≥ 38º C with upper respiratory tract manifestations, generalized bone ache with or without gastrointestinal symptoms as diarrhea.
* Chest CT with signs suggestive of COVID-19.
* Mild and moderate cases of COVID-19 pneumonia with respiratory and hemodynamic stability. - High C reactive protein (CRP).- With or without history of contact with index case who is isolated in a governmental hospital assigned for treatment of patients proved to have RT-PCR positive test for COVID-19
* With or without abnormalities in the total or differential white cell count.
* Welling to sign a fully informed consent.

Exclusion Criteria:

* Severe and critical illness with respiratory failure and/ or hemodynamic instability.
* CT with pleural effusion with or without lung cavitation.
* Other organ failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to clinical recovery | 7 days
  defined as return of body temperature and relief of cough for more than 72 hours measured in days

SECONDARY OUTCOMES:
Pulmonary recovery status | 7 days
  assessed by Chest CT defined as exacerbated, unchanged, moderately improved (with less than 50% pneumonia resolved) and significantly improved (with more than 50% pneumonia resolved).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed K Elbadrawy, PhD, Principal Investigator — Chest department Mansoura University Hospital
Locations (1):
- Gomhoria Street, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No